CLINICAL TRIAL: NCT02809911
Title: A Randomized, Sham-Controlled, Double-Blind, Crossover Study to Evaluate PEMF Therapy on Pain Sensitivity to Different Qualities of Experimentally Induced Pain in Subjects With Painful Peripheral Diabetic Neuropathy
Brief Title: A Study to Evaluate PEMF Therapy on Experimentally Inducted Pain in Subjects With Painful Peripheral Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RBI.2016.002
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2016-10

CONDITIONS: Painful Peripheral Diabetic Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham of Provant (Other): Sham of Provant Therapy System
  Interventions: Device: Provant
- Active Provant (Other): Active Provant Treatment
  Interventions: Device: Provant

INTERVENTIONS:
Device: Provant

SUMMARY:
Evaluate the effectiveness of the Provant Therapy System compared to sham on pain sensitivity and nervous system response to various qualities of experimentally induced pain in the upper and lower extremities of subjects with painful peripheral diabetic neuropathy.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, sham-controlled crossover clinical trial conducted on subjects with painful peripheral diabetic neuropathy. Eligible subjects will include those between 22 and 80 years of age with Type 2 diabetes having persistent pain, numbness, tingling, and/or burning in at least one foot. Pain threshold, tolerance to thermal stimuli and pressure response to the induced pain stimuli will be measured at three time points using five standardized experimental pain measures: baseline, after a single 30 minute treatment with active PEMF or sham treatment and after a second 30 minute treatment with active PEMF or sham treatment. Eligible subjects with painful peripheral diabetic neuropathy will undergo Diabetic Screening (Nerve Conduction Velocity, Skin Perfusion Pressure, Ankle-Brachial Index, and Vibratory Testing) in the index foot prior to randomization. Following the Diabetic Screening tests, subjects will return to the research center for the Enrollment/Randomization Visit and complete measures of pain by completing the Brief Pain Inventory (BPI) and functional assessments. Subjects will then be randomly assigned to one of the two groups; control (sham) or experimental (active) device by a research assistant blinded to the device status. Patients will also be randomly assigned to the sequence order of experimental induced pain tests. The ischemic pain testing (SMET) will always be conducted last. Patients will return to the research center within 7 days after the Enrollment/Randomization Visit where they will be crossed over to the other treatment assignment and be randomly assigned to the sequence order of experimental induced pain tests on the same extremity as previously randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is greater than or equal to 22 years and less than 80 years of age.
2. Subject has documented Type 2 diabetes.
3. Subject's BMI ≤ 38.
4. Subject has peripheral diabetic neuropathy with pain, numbness, tingling, and/or burning in at least one foot.
5. Subject is in pain Phase 2, 3, or 4 (Appendix B).
6. Subject is willing to forego smoking during the Enrollment Visit and Visit 3 (Crossover) for 4 hours prior to and through the duration of testing (~5 hours).
7. Subject is willing and able to give written informed consent and to comply with all parts of the study protocol.
8. Female subjects must be post-menopausal, surgically sterile, abstinent, or practicing (or agree to practice) an effective method of birth control if they are sexually active for the duration of the study. (Effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier methods, and/or male partner sterilization).
9. Subject is able to eat in the morning prior to the induced pain tests and provide a meal/snacks for themselves during the day to maintain blood sugar levels.

Exclusion Criteria:

1. Subject has current pain other than their painful peripheral diabetic neuropathy.
2. Subject has a concomitant medical condition that, in the opinion of the investigator, would confound the ability to conduct induced pain testing in the upper and lower extremities.
3. Subject has taken prescription opioids for their pain within 30 days of the Screening Visit or 6 weeks of Screening for long acting medications.
4. Subject has used topical capsaicin within 30 days of the Screening Visit.
5. Subject has Type 1 diabetes.
6. Subject is in pain Phase 1 or 5 (Appendix B).
7. Subject has an active, open ulcer on either lower extremity of arterial, venous or mixed disease origin.
8. Subject has peripheral arterial disease as determined by an Ankle-Brachial Index (ABI) of <0.5 or > 1.4. See Appendix C for details on obtaining the ABI.
9. Subject has venous insufficiency classified by the Venous Insufficiency Classification System (CEAP) of grade C6. See Appendix D for description of the venous insufficiency grading.
10. Subject has an unhealed surgery on the legs, feet, arms or hands.
11. Subject has smoked within 4 hours of the Screening Visit.
12. Subject has received any investigational drug or device within 30 days or 5 half-lives of the drug, whichever is longer, prior to the Screening Visit or is enrolled in another clinical trial.
13. Subject has used systemic corticosteroids within 2 months of the Screening Visit.
14. Subject has a history of a solid tumor that is not in complete remission for greater than 2 years other than successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin in the treatment area.
15. Subject has a serious psychosocial co-morbidity.
16. Subject has a self-reported history of drug or alcohol abuse, within one year prior to the Screening Visit.
17. Subject has an implanted pacemaker, defibrillator, neurostimulator, spinal cord stimulator, bone stimulator, cochlear implant, or other implanted device with an implanted metal lead(s).
18. Subject is currently pregnant.
19. Subject has been previously treated with the PROVANT Therapy System within 30 days of the Enrollment Visit.
20. Subject is unwilling or unable to follow study instructions.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sun Research Institute, San Antonio, Texas
  - Multi-Phase Trials, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to an error in the randomization for this study, results are based upon data only for the Initial Treatment population (those subjects treated with either active or sham at the Enrollment Visit). Data from the cross-over was not included since the majority of subjects were not crossed-over to the other treatment.
Groups:
- Sham of Provant: Sham of Provant Therapy System
  Provant
- Active Provant: Active Provant Treatment
  Provant
Period: Overall Study
Arm/Group | Sham of Provant | Active Provant
Started | 22 (This is the Initial Treatment Population (subjects that started the Enrollment Visit / Visit 2)) | 19 (This is the Initial Treatment Population (subjects that started the Enrollment Visit / Visit 2))
Completed | 22 (This is the Initial Treatment Population (subjects that completed the Enrollment Visit / Visit 2)) | 19 (This is the Initial Treatment Population (subjects that completed the Enrollment Visit / Visit 2))
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sham of Provant: Sham of Provant Therapy System
  Due to an error in the randomization for this study, results are based upon data only for the Initial Treatment population (those subjects treated with either active or sham at the Enrollment Visit). Data from the cross-over was not included since the majority of subjects were not crossed-over to the other treatment.
- Active Provant: Active Provant Treatment
  Due to an error in the randomization for this study, results are based upon data only for the Initial Treatment population (those subjects treated with either active or sham at the Enrollment Visit). Data from the cross-over was not included since the majority of subjects were not crossed-over to the other treatment.
- Total: Total of all reporting groups
Arm/Group | Sham of Provant | Active Provant | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12.14) | 63.8 (12.38) | 63.4 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 18
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 19 | 16 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 41
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.6 (4.89) | 29.4 (5.17) | 30 (5)

OUTCOME MEASURES:

1. Primary Outcome: Upper Extremity - Pain Sensitivity to Various Experimentally Induced Pain Stimuli
Description: Response data by induced pain stimuli after the initial treatment with the study device in the upper extremity. The stimuli / test was determined to either favor sham or favor Provant Therapy. This included a total of 20 stimuli/tests (comparing pre-treatment to post initial treatment results) as follows: Cuff Pain Threshold (greater decrease favored), Cuff Pain Tolerance (smaller increase favored), Cuff Pressure Threshold (greater decrease favored), Pressure Tolerance (greater increase favored), Mechanical Pain Threshold (greater decrease favored), Biothesiomety (greater decrease favored) on the forearm, palm, thumb, index finger, middle finger, ring finger and pinky finger, Heat Tolerance (greater decrease favored), Cold Tolerance (greater decrease favored), Pain (greater increase favored), Time to Pain (greater increase favored), Pain Tolerance Grip Strength (greater increase favored) and Final Pain (greater decrease favored).
Time Frame: 4 weeks
Population: Due to an error in the randomization for this study, results are based upon data only for the Initial Treatment population (those subjects treated with either active or sham at the Enrollment Visit). Data from the cross-over was not included since the majority of subjects were not crossed-over to the other treatment.
Measure: Number; unit: Number of tests favoring arm/group
Arm/Group | Sham of Provant | Active Provant
Number analyzed (Participants) | 22 | 19
Number of tests favoring arm/group | 6 | 14

2. Primary Outcome: Lower Extremity - Pain Sensitivity to Various Experimentally Induced Pain Stimuli
Description: Response data by induced pain stimuli after the initial treatment with the study device in the upper extremity. The stimuli / test was determined to either favor sham or favor Provant Therapy. This included a total of 20 stimuli/tests (comparing pre-treatment to post initial treatment results) as follows: Cuff Pain Threshold (greater decrease favored), Cuff Pain Tolerance (smaller increase favored), Cuff Pressure Threshold (greater decrease favored), Pressure Tolerance (greater increase favored), Mechanical Pain Threshold (greater decrease favored), Biothesiomety (greater decrease favored) on the forearm, palm, thumb, index finger, middle finger, ring finger and pinky finger, Heat Tolerance (greater decrease favored), Cold Tolerance (greater decrease favored), Pain (greater increase favored), Time to Pain (greater increase favored), Pain Tolerance Grip Strength (greater increase favored) and Final Pain (greater decrease favored). .
Time Frame: 4 weeks
Population: Includes subjects in the Initial Treatment Group (Those subjects treated with either Provant or Sham at the Enrollment Visit)
Measure: Number; unit: Number of tests favoring arm/group
Arm/Group | Sham of Provant | Active Provant
Number analyzed (Participants) | 22 | 19
Number of tests favoring arm/group | 16 | 4

ADVERSE EVENTS:
Arm/Group | Sham of Provant | Active Provant
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 0/22 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication Rights. Independent analysis and/or publication of data is not permitted without the prior written consent of the sponsor. Such consent may be contingent on sponsor review and approval of any proposed analysis and manuscript. Institution will retain the right to review and analyze the database created from this study for its own scientific purposes so long as such scientific purposes are non-commercial in nature.